CLINICAL TRIAL: NCT05030220
Title: Association Between Serum Testosterone Levels and Cutibacterium Culture Positivity During Shoulder Arthroplasty
Brief Title: Testosterone Levels and Cutibacterium
Status: Recruiting | Type: Observational
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Jason Hsu, Associate Professor, School of Medicine, University of Washington
Other Study IDs: STUDY00009200
Record Dates: First submitted 2021-05-07; First posted 2021-09-01 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Arthroplasty, Replacement, Shoulder
Keywords: Testosterone; Cutibacterium; Shoulder Arthroplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Phase 1: 51 subjects with serum levels of testosterone, free testosterone, and sex hormone binding globulin as well as the SpCuV from the cultures obtained in clinic, immediately pre-operative skin cultures, and incised wound cultures.
- Phase 2: Subjects enrolled to help determine if preoperative serum testosterone levels are associated with risk for shoulder PJI in patients undergoing primary shoulder arthroplasty and if preoperative serum testosterone levels are predictive of bacterial load of deep tissue cultures taken at the time of revision shoulder arthroplasty in patients undergoing primary shoulder arthroplasty.

SUMMARY:
Phase 1: In 51 patients undergoing shoulder arthroplasties, total serum testosterone, free testosterone and sex hormone binding globulin levels obtained in the clinic before surgery were correlated with the levels of Cutibacterium on the skin in clinic, in the operating room prior to surgery, and in the skin incision.

Phase 2: The investigators wish to determine if preoperative serum testosterone levels are associated with risk for shoulder PJI (periprosthetic joint infection) in patients undergoing primary shoulder arthroplasty. Also to determine if preoperative serum testosterone levels are predictive of bacterial load of deep tissue cultures taken at the time of revision shoulder arthroplasty in patients undergoing primary shoulder arthroplasty.

DETAILED DESCRIPTION:
Phase 1: 51 patients having elective shoulder arthroplasty were offered the opportunity to participate, consented and enrolled in this prospective clinical cohort study.

At a preoperative clinic visit, basic demographic information was collected along with the patient's response to a question about taking supplemental testosterone. A swab of the unprepared skin over the area of the intended surgical incision was obtained and sent for culture. At this clinic visit, a sample of the patient's blood was also obtained and submitted to our clinical laboratory for the levels of total serum testosterone, sec hormone binding globulin (SHBG), and free testosterone.

Immediately before surgery, another swab of the unprepared skin over the area of the intended surgical incision was once again obtained and sent for culture. After incision, a swab of the freshly incised dermis was obtained and sent for culture.

All 3 swabs that were obtained were observed for 21 days. The investigators analyzed the cultures to determine the presence and load of bacteria using a semiquantitative method, known as the Cutibacterium specimen value (SpCuV)

Phase 2: This phase will also involve a onetime pre-operative testosterone serum test. If the subject consents to participate, this additional sample of blood will be collected for a testosterone serum test during the routine pre-operative blood draw that all patients have before a shoulder arthroplasty regardless of research participation. The investigators will include cultures such as skin swabs taken at pre-operative clinic appointments, skin swabs taken at the time of surgery, incision swabs taken at the time of surgery, and discarded tissue from surgery using our standard protocol for specimens. For this study's outcome measures, the investigators will record the culture results from those clinical specimens and compare them to the testosterone serum test. Some subjects may also be a part of a long term follow-up study and the follow-up data (self-reported outcome measures, etc.) from that study will be included for analysis for those patients.

ELIGIBILITY:
Phase 1 Inclusion Criteria:

* Patients having elective shoulder arthroplasty

Phase 1 Exclusion Criteria:

* history of shoulder septic arthritis
* antibiotic use within 3 months prior to surgery
* recent treatment for acne
* Lacked fluency in English

Phase 2 Inclusion Criteria:

* Patients having elective shoulder arthroplasty

Phase 2 Exclusion Criteria:

* Lacked fluency in English

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Phase 1 and 2: Subjects will be adult patients who present to the UWMC Bone & Joint Center for pre-operative appointments for elective shoulder arthroplasty.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Serum testosterone | At pre-operative clinic appointment, typically within 30 days prior to surgery
Free testosterone | At pre-operative clinic appointment, typically within 30 days prior to surgery
sex hormone binding globulin | At pre-operative clinic appointment, typically within 30 days prior to surgery
Cutibacterium specimen value | Skin swab at pre-operative clinic appointment, typically within 30 days prior to surgery
Cutibacterium specimen value | Skin swab immediately pre-operative
Cutibacterium specimen value | Freshly incised dermis of surgical wound
Preoperative serum testosterone levels are associated with risk for shoulder PJI in patients undergoing primary shoulder arthroplasty. | Up to 20 years after surgery
Preoperative serum testosterone levels are predictive of bacterial load of deep tissue cultures taken at the time of revision shoulder arthroplasty in patients undergoing primary shoulder arthroplasty | 21 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jason E Hsu, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No